CLINICAL TRIAL: NCT06735833
Title: Feasibility Study to Evaluate the Initial Safety and Effectiveness of TRUFILL n-BCA Liquid Embolic System in Middle Meningeal Artery Embolization for the Preventive Treatment of Refractory Chronic Migraine
Brief Title: MMA Embolization for Refractory Chronic Migraine
Acronym: Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CNV202302; CNV202302 (Other: Cerenovus, Part of DePuy Synthes Products, Inc)
Record Dates: First submitted 2024-12-04; First posted 2024-12-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, feasibility study in which up to 50 subjects will be consented to achieve a total of 30 subjects treated with TRUFILL n-BCA bilateral middle meningeal artery (MMA) embolization for the treatment of refractory chronic migraine in up to 5 US centers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Middle Meningeal Artery embolization — Bilateral middle meningeal artery embolization using TRUFILL n-BCA liquid embolic system

SUMMARY:
This is a prospective, multi-center, feasibility study to investigate safety and effectiveness of TRUFILL n-BCA liquid embolic system in bilateral middle meningeal artery (MMA) embolization for the treatment of refractory chronic migraine.

ELIGIBILITY:
Participant Inclusion Criteria, Candidates for this study must meet ALL the following inclusion criteria:

1. Patient is between 18 and 65 years of age (inclusive) at the time of consent.
2. Age of onset of Chronic Migraine ≤ 64 years.
3. Age of onset of migraine diagnosis < 50 years.
4. Patient has a current diagnosis of refractory migraine.
5. Patient has a current diagnosis of Chronic migraine.

Participant Exclusion Criteria, Candidates will be excluded from participation if ANY of the following apply:

1. Patients with a history for the last 2 years of other types of headache. 2. Patients with diagnosis of hemiplegic migraine or migrainous infarct. 5. Patients with current regular use of Opioids, Cannabis, Medical Marijuana, etc.

6. Women who are pregnant, lactating, or who are of childbearing age. 7. Current involvement in an investigational (drug, device, etc.) clinical trial that may confound study endpoints. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible. Sponsor approval is required.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2028-12-25 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline, in number of migraine days | over 28 days

SECONDARY OUTCOMES:
Change from baseline in migraine days frequency | 3 months and 6 months

OTHER OUTCOMES:
Serious Adverse events | At 4 weeks, 3 months, 6 months and 1 Year

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Mount Sinai, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Semmes Murphey Foundation, Memphis, Tennessee
  - West Virginia University, Morgantown, West Virginia